CLINICAL TRIAL: NCT06254599
Title: A Phase III Study to Evaluate and Compare the Efficacy and Safety of SY-3505 Versus Crizotinib in Treatment-Naive Patients With Anaplastic Lymphoma Kinase (ALK)-Positive Advanced Non-Small Cell Lung Cancer
Brief Title: A Study Of SY-3505 Versus Crizotinib In First Line Treatment Of Patients With ALK-Positive NSCLC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shouyao Holdings (Beijing) Co. LTD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-3505-III-01
Record Dates: First submitted 2024-02-01; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: SY-3505; Anaplastic lymphoma kinase; Non-small Cell Lung Cancer; Third-generation ALK tyrosine kinase inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SY-3505 (Experimental): SY-3505, single agent, 600 mg oral capsules, QD, continuously
  Interventions: Drug: SY-3505 Capsules
- Crizotinib (Active Comparator): Crizotinib, single agent, 250 mg oral capsules, BID, continuously
  Interventions: Drug: Crizotinib Capsules

INTERVENTIONS:
Drug: SY-3505 Capsules — A third-generation ALK tyrosine kinase inhibitor
  Other Names: CT-3505; Ficonalkib
  Arms: SY-3505
Drug: Crizotinib Capsules — An oral ALK tyrosine kinase inhibitor
  Other Names: Xalkori
  Arms: Crizotinib

SUMMARY:
A phase 3 study to evaluate the efficacy and safety of SY-3505 vs. crizotinib in patients with ALK-positive non-small cell lung cancer who had not received prior systemic therapy.

DETAILED DESCRIPTION:
This is a multicenter, randomized controlled phase III trial to evaluate the efficacy and safety of SY-3505 capsule vs. crizotinib capsule in treatment-naive patients with ALK-positive NSCLC.

Participants will be randomized in a 2:1 ratio to receive SY-3505, 600 milligrams (mg) orally once daily (QD), or crizotinib, 250 mg orally twice daily (BID). Participants will receive treatment until disease progression, unacceptable toxicity, withdrawal of consent, or death.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the informed consent form (ICF), age is ≥ 18 years.
2. Histologically or cytologically diagnosed with stage IV or stage IIIB and IIIC NSCLC that cannot be cured by surgery or radiotherapy (as per the 8th edition of the International Association for the Study of Lung Cancer [IASLC] Lung Cancer Staging).
3. No prior systemic anti-tumor therapy for NSCLC, including but not limited to systemic chemotherapy, ALK-TKI, immunotherapy, and biologic therapy, etc. [1. Patients assessed by the investigator as not having received "adequate" systemic anti-tumor therapy (such as having received up to 1 prior chemotherapy regimen, etc.), and 2. Patients who have received neoadjuvant or adjuvant therapy, with the last treatment at least 6 months before randomization, are allowed to be included].
4. The tumor tissue or blood sample of the patient meets one of the following two criteria: a. Previously confirmed by a local laboratory as ALK fusion-positive (patients included based on previously confirmed ALK fusion-positive test results should provide tumor tissue [available archived samples or fresh biopsy samples] that meets the requirements as much as possible after signing the ICF and before the first dose for central laboratory ALK fusion positive reconfirmation based on study progression needs). b. In the absence of a previous ALK fusion positive test report, a tumor tissue (available archived samples or fresh biopsy samples) or blood sample meeting the requirements must be provided, and the sample is confirmed as ALK fusion positive in the designated center laboratory by the sponsor.
5. At least one extra-cranial target lesion that meets the RECIST v 1.1 criteria definition; for lesions previously treated with radiotherapy, only when the lesion shows clear progression after radiotherapy can it be considered a target lesion.
6. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-2.
7. Expected survival time of ≥ 3 months.
8. Before the first dose, the adverse events (AEs) related to previous anti-tumor therapy have recovered to Grade ≤ 1 as defined by NCI-CTCAE v 5.0 (excluding toxicities judged by the investigator to have no safety risks, such as alopecia, Grade 2 peripheral neuropathy related to previous platinum-based treatment, etc.).
9. Organ function levels must meet the following requirements (supportive treatment that affects the following results has not been received within 7 days before the test):

   * Bone marrow function: Absolute neutrophil count (ANC) ≥ 1.0×10^9/L, platelets (PLT) ≥ 75×10^9/L, hemoglobin (Hb) ≥ 90g/L;
   * Liver function: In the absence of liver metastasis, serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) both ≤ 2.5× the upper limit of normal (ULN), and serum total bilirubin (TBIL) ≤ 1.5× ULN; with liver metastasis, AST and ALT both ≤ 5.0× ULN, and TBIL ≤ 3× ULN;
   * Renal function: Creatinine clearance rate (Ccr) ≥ 50 mL/min (according to the Cockcroft and Gault formula);
   * Coagulation function: International normalized ratio (INR) and prothrombin time (PT) ≤ 1.5× ULN (except for patients receiving anticoagulant therapy).
10. Able to swallow pills and able to comply with the visits and related procedures as specified in the protocol.
11. Fertile subjects agree to use effective contraceptive measures during the entire study period and for at least 3 months after the last dose

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible to participate in this study:

1. Carrying known major driver gene mutations other than ALK, such as EGFR, MET, RET, ROS1, NTRK, etc. (patients with co-mutations can discuss with the investigator whether they can be included).
2. History of allergy to any component or excipient of SY-3505 capsules or crizotinib capsules.
3. Concurrent primary malignancies, with the following exceptions: cured and not relapsed malignant tumors within 2 years before screening, and cured basal cell carcinoma or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or carcinoma in situ of the breast.
4. Presence of symptomatic primary central nervous system (CNS) tumors, symptomatic CNS metastases, leptomeningeal carcinomatosis, or untreated spinal cord compression. Exception: Patients with stable CNS conditions (no evidence of progression on imaging examinations for at least 4 weeks before the first dose and all neurological symptoms have returned to baseline), no evidence of new or enlarged brain metastases, no CNS surgery or radiotherapy within 4 weeks before the first dose, no stereotactic radiosurgery (SRS) within 2 weeks, and discontinuation or stable dose of steroids within 2 weeks (this exception does not include carcinomatous meningitis, which should be excluded regardless of its clinical status).
5. Concomitant symptoms or diseases before the first dose that are poorly controlled even after optimal treatment (chronic diseases do not require screening):

   * Uncontrolled active systemic bacterial, viral, or fungal infections;
   * Pleural effusion, ascites, or pericardial effusion poorly controlled after intervention (poorly controlled indicates significant increase in effusion within 2 weeks after drainage, with significant symptoms requiring re-puncture or other interventions);
   * Poorly controlled diabetes (fasting blood glucose ≥ 11.1mmol/L and/or HbA1c ≥ 8%);
   * Symptomatic hyperthyroidism or hypothyroidism that is not controlled according to the investigator's assessment;
   * Clinically significant electrolyte disturbances evaluated by the investigator (such as hypocalcemia, hypomagnesemia, or hypokalemia);
   * Clinically significant active gastrointestinal diseases, including active ulcerative colitis, Crohn's disease, gastrointestinal ulcers, or previous surgical procedures that may significantly affect drug absorption.
6. Presence of severe cardiovascular diseases/abnormalities, meeting any of the following:

   * Fridericia-corrected QT interval (QTcF) > 470 msec (females) or 450 msec (males) during screening (if QTcF prolongation suspected to be drug-induced is assessed as safe and controllable by the investigator, the patient can be included after correction with medication);
   * Left ventricular ejection fraction (LVEF) < 50%;
   * Myocardial infarction or unstable angina within 6 months before the first dose or clinically significant uncontrolled arrhythmias, including bradycardias that may lead to QTcF prolongation (such as type II second-degree or third-degree atrioventricular block);
   * Classified as New York Heart Association (NYHA) class III or IV congestive heart failure;
   * Poorly controlled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg), history of unstable hypertension, or poor compliance with antihypertensive treatment.
7. Active viral infections or history of the following:

   * Hepatitis B during screening (positive results for hepatitis B surface antigen [HBsAg] and/or hepatitis B core antibody [HBcAb] with HBV-DNA ≥2×103 IU/mL; patients whose HBV-DNA levels drop to below 2×103 IU/mL after regular antiviral treatment can be included), or active hepatitis C (HCV RNA > central detection upper limit of normal [ULN]);
   * Human immunodeficiency virus (HIV) positive during screening, or known history of other immunodeficiency diseases, or receiving long-term systemic corticosteroid therapy (daily dose of prednisone exceeding 10 mg or equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose;
   * History of organ transplantation, hematopoietic stem cell, or bone marrow transplantation.
8. Other lung diseases requiring systemic treatment or severe lung diseases, such as active pulmonary tuberculosis, interstitial lung disease, etc., which, in the investigator's judgment, may affect the interpretation of the study results or put the patient at high risk.
9. Use of or inability to stop using the following CYP3A4 potent inhibitors or inducers within 2 weeks before the first dose during the study. CYP3A4 potent inhibitors: Atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, grapefruit (juice); CYP3A4 potent inducers: Carbamazepine, phenobarbital, phenytoin, rifampicin, St. John's wort, rifabutin.
10. Underwent radiotherapy within 2 weeks before the first dose or experienced radiation-related toxicities requiring corticosteroid therapy.
11. Used Chinese herbal medicine or preparations with indications for anti-tumor therapy or tumor adjuvant therapy within 2 weeks before the first dose.
12. Underwent major surgery within 4 weeks before the first dose (major surgery defined as surgery with a grade ≥3, excluding central venous catheter placement, tumor biopsy, and gastric tube insertion) or experienced significant trauma and has not fully recovered.
13. Participated in other clinical trials within 4 weeks before the first dose (Note: Except for those who did not use investigational drugs or investigational medical devices; those who stopped treatment in other clinical trials and only underwent follow-up for survival period).
14. Received lung radiotherapy >30 Gy within 6 months before the first dose.
15. Experienced severe arterial/venous thrombotic events within 1 year before the first dose (such as cerebrovascular accident [including transient ischemic attack], deep vein thrombosis, pulmonary embolism) and judged by the investigator as not suitable for participation in this trial, or has a significant bleeding tendency within 30 days before the first dose, or judged by the investigator to have a risk of significant gastrointestinal bleeding, etc.
16. Pregnancy (screening pregnancy test result for women of childbearing age must be negative) or breastfeeding women.
17. Other situations deemed unsuitable for participation in this clinical trial by the investigator, such as other severe acute or chronic diseases that may increase the patient's related risks in the study or laboratory abnormalities that may interfere with the interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by independent radiology review (IRC) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1) criteria. | Up to 2 years
  PFS was defined as the time from randomization to the date of the first documentation of progressive disease as assessed by the independent radiologist or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
Progression-free survival (PFS) assessed by investigator based on RECIST v1.1 criteria. | Up to 2 years
  PFS was defined as the time from randomization to the date of the first documentation of progressive disease as assessed by the independent radiologist or death due to any cause, whichever occurred first.
Objective Response Rate (ORR) assessed by IRC and investigator | Up to 2 years
  ORR is defined the percentage of the participants who have achieved complete response (CR) or partial response (PR) per IRC and investigator based on RECIST v1.1 after the initiation of study treatment.
Disease Control Rate (DCR) assessed by IRC and investigator | Up to 2 years
  DCR is defined the percentage of the participants who have achieved an objective response (CR or PR) or stable disease (SD) per IRC and investigator based on RECIST v1.1 after the initiation of study treatment.
Duration of Response (DoR) assessed by IRC and investigator | Up to 2 years
  DoR is defined as the time from the first occurrence of an objective response (CR or PR), based on RECIST v1.1 to first documented disease progression or death.
Intracranial Objective Response Rate (IC-ORR) assessed by IRC and investigator | Up to 2 years
  IC-ORR is defined as the proportion of patients with intracranial target lesions that are measurable at baseline who achieve an objective response (CR or PR) according to RECIST 1.1 and Revised Assessment in Neuro Oncology (RANO) criteria.
Intracranial Disease Control Rate (IC-DCR) assessed by IRC and investigator | Up to 2 years
  IC-DCR is defined as the proportion of patients with intracranial target lesions that are measurable at baseline who achieve an objective response (CR or PR) or SD according to RECIST 1.1 and Revised Assessment in Neuro Oncology (RANO) criteria.
Intracranial Duration of Response (IC-DoR) assessed by IRC and investigator | Up to 2 years
  IC-DoR was defined as time from documentation of intracranial response (CR or PR) to intracranial disease progression or death.
Overall Survival (OS) | Up to 2 years
  OS is defined as the time interval from the date of the first dose of the study treatment until death due to any cause. It will be censored on the date of last contact for those participants who are alive.

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Sun, Study Director — Shouyao Holdings (Beijing) Co. LTD
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China